CLINICAL TRIAL: NCT04117555
Title: Assessment of Pupil Light Reflex in Patients With Parkinson Disease in Comparison to Healthy Subjects.
Brief Title: Assessment of Pupil Light Responses in Patients With Parkinson Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Sharon Hassin, Prof., Sheba Medical Center
Other Study IDs: 5956-19
Record Dates: First submitted 2019-09-18; First posted 2019-10-07 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Diagnostic Test: Pupillometry
  Interventions: Diagnostic Test: Pupil response to light stimuli
- Parkinson patients: Diagnostic Test: Pupillometry
  Interventions: Diagnostic Test: Pupil response to light stimuli

INTERVENTIONS:
Diagnostic Test: Pupil response to light stimuli — Objective and accurate measurement of pupillary responses to light stimuli

SUMMARY:
Parkinson diseases (PD) is the second most common degenerative disease of the central nervous system. The development of early diagnostic biomarkers may help identify at-risk individuals and allow precocious interventions at the onset of disease and more precise monitoring of therapies that may slow disease progression.

Proof of concept studies indicated significant differences in pupil light response between PD patients and healthy controls. The feasibility of using pupillometry for assesment of PD will be examined.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria

  1. Age 30-75 years old
  2. Signed written informed consent
  3. Gender: Both (Male and Female)
  4. Pupillary reflex to light.
  5. Clear ocular media

Patients' Inclusion Criteria:

Patients with clinical presentations of the neurodegenerative forms of parkinsonism (bradykinesia, extrapyramidal rigidity, tremor, postural instability and gait disturbance) including: idiopathic Parkinson disease (PD), Lewy body disease (LBD), progressive supranuclear palsy (PSP), multiple system atrophy (MSA), corticobasal degeneration (CBD) and secondary parkinsonisms.

Control group- inclusion criteria

1. Normal eye examination
2. Best-corrected visual acuity (BCVA) of 20/20
3. Normal color vision test (Farnsworth/Lanthon D-15 Test)
4. No present ocular disease
5. No past ocular disease or surgery within last 6 months
6. No use of any topical or systemic medications that could adversely influence efferent pupil movements
7. Normal 24-2 Humphrey visual field and

   * Short duration (≤10 minutes)
   * Minimal fixation losses, False positive errors and False negative errors (less than 30% for each one of reliability indices)

Exclusion Criteria:

1. Diagnosis of dementia.
2. Cognitive decline that may impair obtaining informed consent.
3. Tremor or dyskinesia that could interfere with ophthalmic evaluation
4. History of past (last 3 months) or present ocular disease or ocular surgery
5. Use of any topical or systemic medications that could adversely influence pupillary reflex
6. Psychiatric illness, active psychosis.
7. Previous neurosurgical interventions, including stereotactic neurosurgical procedures.
8. Past or current strokes or brain injury and other brain disorders (except PD/parkinsonism for patient group)
9. Anti-dopaminergic drugs.
10. Intolerance to gonioscopy, slit lamp examination, Goldmann applanation tomometry or other schedule study procedure.
11. Visual media opacity including cloudy corneas.
12. Any condition preventing accurate measurement or examination of the pupil.

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: One hundred Parkinson patients or patients with parkinsonism and 100 age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pupillometry | 1 day
  Pupil response to light stimuli

SECONDARY OUTCOMES:
Best corrected visual acuity | 1day
  Visual Acuity
Color vision | 1 day
  Color vision by Farnsworth/Lanthon D-15 Test
Humphrey 24-2 perimetry | 1 day
  Visual field will be assessed by Humphrey 24-2 perimetry
Spcetral Domain Optical Coherence Tomography (SD-OCT) | 1 day
  Optic nerve and retinal structure will be assessed by SD-OCT
visual evoked potential | 1 day
  Occipital cortex function will be assessed by visual evoked potential (VEP)
Change from baseline Pupillometry at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline in pupil response to light stimuli at 1 year
Change from baseline best corrected visual acuity at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline visual acuity at 1 year
Change from baseline color vision at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline color vision by Farnsworth/Lanthon D-15 at 1 year
Change from baseline Humphrey 24-2 at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline Humphrey 24-2 visual field at 1 year
Change from baseline SD-OCT at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline optic nerve and retinal structure by SD-OCTat 1 year
Change from baseline visual evoked potential at 1 year | Single visit: 1 day, 1 year after baseline testing
  Change from baseline occipital cortex function by visual evoked potential testing to at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hassin-Baer, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Goldschleger Eye Research Institute, Sheba Medical Center,, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No